CLINICAL TRIAL: NCT00529789
Title: F1J-MC-HMFN (a) An Open-Label Study of Tolerability, Safety, and Pharmacokinetics of Duloxetine in the Treatment of Children and Adolescents With Major Depressive Disorder
Brief Title: Open-Label Study of Duloxetine in the Treatment of Children and Adolescents With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11664; F1J-MC-HMFN (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2009-12-09 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental)
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — 20 - 120 milligrams (mg) every day, once-daily (QD), by mouth (PO) for 30 weeks; If patient is ≤40 kilograms (kg), initial dose is 20 mg, then titrated up. If patient is >40 kg, initial dose is 30 mg, then titrated up.
  Other Names: LY248686; Cymbalta

SUMMARY:
The primary purpose of your participation in this study is to help answer the following research question, and not to provide you treatment for your condition. Whether duloxetine once daily orally is tolerated and safe, in children (aged 7 through 11 years) and adolescents (aged 12 through 17 years) with Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male / Female outpatients 7 to 17 years of age diagnosed with Major Depressive Disorder (MDD). (Must have a Children's Depression Rating Scale-Revised [CDRS-R] with a total score greater than or equal to 40 at Visit 1, Visit 2, and Visit 3 and a Clinical Global Impressions of Severity [CGI-Severity] rating of greater than or equal to 4 at Visit 1, Visit 2, and Visit 3.)
* Female patients must test negative on a pregnancy at visit 1.

Exclusion Criteria:

* Have a serious or unstable medical illness, psychological condition, clinically significant laboratory or electrocardiogram (ECG) result, hypersensitivity to duloxetine, or to its inactive ingredients, frequent or severe allergic reactions to multiple medications, uncontrolled narrow-angle glaucoma, acute liver injury (for example, hepatitis) or severe cirrhosis (Child-Pugh Class C) that in the opinion of the investigator would compromise participation in the study or be likely to lead to hospitalization during the course of the study.
* Have a current or previous diagnosis of bipolar disorder, psychotic depression, schizophrenia or other psychotic disorder, anorexia, bulimia, obsessive compulsive disorder, pervasive development disorder or borderline personality disorder, as determined by the investigator.
* Have a significant suicide attempt within 1 year of Visit 1 or have a score of 5 or greater on Item 13 (Suicidal Ideation) on the CDRS-R at Visit 1, Visit 2, or Visit 3, or are currently at risk of suicide in the opinion of the investigator.
* Have a weight less than 20 kg at any Screening Phase visit.
* Have previous exposure to duloxetine
* Female patients who are either pregnant, nursing or have recently given birth.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern Standard time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- United States (22):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dothan, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chandler, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Centro, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eagle, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terre Haute, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Kisco, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Jackson, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herndon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midlothian, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period I was a 2-week Screening/Washout Phase. Period II was a 10-week Dose-Titrating with Pharmacokinetic Sampling Phase. Period III was an 8-week Safety and Tolerability Phase. Period IV was a 3-month Extended Safety and Tolerability Phase. Period V was a 2-week Taper Phase. Results presented are for combined Periods II/III and Period IV.
Period: Study Period II/III
Arm/Group | Duloxetine
Started | 72
Completed | 48
Not Completed | 24
Not completed — Parent/Caregiver Decision | 9
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 3
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 3
Period: Study Period IV
Arm/Group | Duloxetine
Started | 48
Completed | 42 (Includes 1 patient who withdrew at last visit; didn't enter Taper; however received 30 weeks of drug)
Not Completed | 6
Not completed — Parent/Caregiver Decision | 1
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 12.5 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 72
Race/Ethnicity [Number; unit: participants]
  African | 17
  Caucasian | 42
  East Asian | 1
  Hispanic | 11
  Native American | 1
Tobacco Use [Number; unit: participants] — Tobacco use was based on cotinine level.
  participants
    No | 70
    Yes | 1
    Not Available | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 23.7 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Emergence of Suicidal Ideation During Period II/III
Description: Emergence of Any Suicidal Ideation: Item 13 of Children's Depression Rating Scale-Revised (CDRS-R) has possible scores of 1 (no thoughts of suicide) to 7 (contemplation of suicide). Emergence of suicidal ideation was defined as an increase in severity of suicidal ideation for those patients who did not have suicidal ideation at baseline (Week 0).
Time Frame: Baseline to 18 weeks
Population: All enrolled patients with data for specified category.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
participants | 2

2. Primary Outcome: Number of Participants With Emergence of Suicidal Ideation During Period IV
Description: as for outcome 1
Time Frame: Week 0 and Between 18 and 30 Weeks
Population: All enrolled patients with data for specified category.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 48
participants | 0

3. Primary Outcome: Number of Participants Experiencing Suicidal Ideation or Suicidal Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS) During Period II/III
Description: The C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. Some questions are yes/no and some are on a scale of 1 (low severity) to 5 (high severity). Completed suicide and non-fatal suicide events are yes/no questions and results presented are the number of participants with these events. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.
Time Frame: Baseline to 18 Weeks
Population: All enrolled patients.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
participants
  Completed suicide | 0
  Non-fatal suicide event | 1
  Worsening of Suicidal Ideation | 1

4. Primary Outcome: Number of Participants Experiencing Suicidal Ideation or Suicidal Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS) During Period IV
Description: as for outcome 3
Time Frame: Between 18 and 30 Weeks
Population: Number of enrolled patients with baseline and post-baseline values in Period IV.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 45
participants
  Completed suicide | 0
  Non-fatal suicide event | 0
  Worsening of Suicidal Ideation | 1

5. Primary Outcome: Number of Participants Meeting Criteria for Potentially Clinically Significant Vital Sign Values at Any Time During Period II/III
Description: Total number of patients with any abnormal post-baseline value, based on all values at scheduled and unscheduled visits. Criteria: High Diastolic Blood Pressure = increase of at least 5 mmHg to a value above the 95th percentile; High Systolic Blood Pressure = increase of at least 5 mmHg to a value above the 95th percentile; High Pulse = increase of at least 25 to a value of at least 110.
Time Frame: Baseline to 18 Weeks
Population: Number of patients with baseline (and none abnormal) and post-baseline values, based on all values at scheduled and unscheduled visits.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
participants
  High Diastolic Blood Pressure | 22
  High Systolic Blood Pressure | 25
  High Pulse | 2

6. Secondary Outcome: Pharmacokinetics: Summary of Observed Duloxetine Plasma Concentrations Stratified by Duloxetine Dose
Description: Plasma samples were obtained at steady state, and approximately 95% of duloxetine concentrations were within the 24 hour dosing interval.
Time Frame: Weeks 2, 4, 6, 8, 10, 14, 18
Population: Number of patients in each duloxetine dose.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Duloxetine Dose - 20 mg: 20 milligrams (mg) every day, once-daily (QD), by mouth (PO); If patient is ≤40kg, initial dose is 20mg, then titrated up.
- Duloxetine Dose - 30 mg: 30 milligrams (mg) every day, once-daily (QD), by mouth (PO); If patient is ≤40kg, initial dose is 20mg, then titrated up. If patient is >40kg, initial dose is 30mg, then titrated up.
- Duloxetine - 60 mg: 60 milligrams (mg) every day, once-daily (QD), by mouth (PO); If patient is ≤40kg, initial dose is 20mg, then titrated up. If patient is >40kg, initial dose is 30mg, then titrated up.
- Duloxetine Dose - 90 mg: 90 milligrams (mg) every day (QD), by mouth (PO); If patient is ≤40kg, initial dose is 20mg, then titrated up. If patient is >40kg, initial dose is 30mg, then titrated up.
- Duloxetine - 120 mg: 120 milligrams (mg) every day, once-daily (QD), by mouth (PO); If patient is ≤40kg, initial dose is 20mg, then titrated up. If patient is >40kg, initial dose is 30mg, then titrated up.
Arm/Group | Duloxetine Dose - 20 mg | Duloxetine Dose - 30 mg | Duloxetine - 60 mg | Duloxetine Dose - 90 mg | Duloxetine - 120 mg
Number analyzed (Participants) | 14 | 53 | 41 | 33 | 19
nanograms per milliliter (ng/mL) | 15.2 (12.0) | 20.8 (21.2) | 41.1 (34.7) | 57.6 (43.2) | 77.6 (54.6)

7. Secondary Outcome: Change From Baseline to 18 Weeks and 30 Weeks in Clinical Global Impressions of Severity Scale (CGI-S)
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Baseline is the same timepoint (Week 0) for both comparisons, but due to differences in number of patients in both periods (II/III vs IV), the baseline values may be slightly different.
Time Frame: Week 0 (Baseline), 18 Weeks, 30 Weeks
Population: 18 Week results are for all enrolled patients with a baseline and at least one non-missing post-baseline value; 30 Week results are for the enrolled patients with a baseline and at least one non-missing post-baseline value in Period IV. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
units on a scale
  18 Week Baseline (n=72) | 4.5 (0.58)
  18 Week Change from Baseline (n=72) | -2.11 (1.17)
  30 Week Baseline (n=45) | 4.5 (0.59)
  30 Week Change from Baseline (n=45) | -2.7 (1.07)

8. Secondary Outcome: Change From Baseline to 18 Weeks and 30 Weeks in Children's Depression Rating Scale-Revised (CDRS-R) Total Score
Description: Measures presence and severity of depression. Consists of 17 items scored on a 1-5 or 1-7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. In general, scores below 20 indicate an absence of depression; scores of 20 or 30 indicate borderline depression; scores of 40 to 60 indicate moderate depression. Baseline is the same timepoint (Week 0) for both comparisons, but due to differences in number of patients in both periods (II/III vs IV), the baseline values may be slightly different.
Time Frame: Week 0 (Baseline), 18 Weeks, 30 Weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
units on a scale
  18 Week Baseline (n=72) | 61.69 (8.98)
  18 Week Change from Baseline (n=72) | -32.11 (12.92)
  30 Week Baseline (n=45) | 61.8 (9.28)
  30 Week Change from Baseline (n=45) | -38.8 (11.14)

9. Primary Outcome: Number of Participants Meeting Criteria for Potentially Clinically Significant Vital Sign Values at Any Time During Period IV
Description: as for outcome 5
Time Frame: Between 18 and 30 Weeks
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 45
participants
  High Diastolic Blood Pressure | 3
  High Systolic Blood Pressure | 1
  High Pulse | 0

10. Primary Outcome: Number of Participants Meeting Criteria for Potentially Clinically Significant (PCS) Laboratory Analyte Values at Any Time During Period II/III
Description: The results shown are for all laboratory analytes where PCS criteria were met, based on criteria used for adult studies. Criteria: High Alanine transaminase (>165 Units/Liter [U/L]); High Creatine Phosphokinase (females: >507 U/L; males:>594 U/L); Low Glucose (<2.498 millimoles/L); Low Hematocrit (females: <0.32; males <0.37); Low Hemoglobin (females <5.896 millimoles/L [mmol/L] iron; males <7.137 mmol/L iron); High Inorganic Phosphorus (>1.776 millimoles/L); Low Leukocyte Count (<2.8 X10^9/L).
Time Frame: Baseline to 18 Weeks
Population: Total number of patients with baseline (and none abnormal) and post-baseline values, based on all values at scheduled and unscheduled visits.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
participants
  High Alanine Transaminase (N=69)) | 1
  High Creatine Phosphokinase (N=69) | 6
  Low Glucose (N=69) | 1
  Low Hematocrit (N=60) | 8
  Low Hemoglobin (N=67) | 1
  High Inorganic Phosphorus (N=62) | 16
  Low Leukocyte Count (N=68) | 1

11. Primary Outcome: Number of Participants Meeting Criteria for Potentially Clinically Significant (PCS) Laboratory Analyte Values at Any Time During Period IV
Description: The results shown are for all laboratory analytes where PCS criteria were met, based on criteria used for adult studies. Criteria: High Alkaline Phosphatase (>420 Units/Liter [U/L]); Low Hematocrit (females <0.32; males <0.37); High Inorganic Phosphorus (>1.776 millimoles/L).
Time Frame: Between 18 and 30 Weeks
Population: Total number of patients with baseline (and none abnormal) and post-baseline values in Period IV, based on all values at scheduled and unscheduled visits.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 48
participants
  High Alkaline Phosphatase (N=42) | 1
  Low Hematocrit (N=39) | 1
  High Inorganic Phosphorus (N=39) | 3

12. Primary Outcome: Number of Participants Meeting Criteria for Potentially Clinically Significant Electrocardiograms at Any Time in Period II/III
Description: Total number of patients with any abnormal post-baseline values, based on all values at scheduled and unscheduled visits. Criteria: High QRS Interval = ≥100 milliseconds (msec); High QTc Bazette's or Fredericia's correction - Female = ≥470 msec; High QTc Bazette's or Fredericia's correction - Male = ≥450 msec.
Time Frame: Baseline to 18 Weeks
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
participants
  High QRS Interval (N=63) | 1
  High QTc Bazette's Correction (N=64) | 2
  High QTc Fredericia's Correction (N=65) | 0

13. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiograms at Any Time in Period IV
Description: as for outcome 12
Time Frame: Between 18 and 30 Weeks
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 48
participants
  High QRS Interval (N=39) | 1
  High QTc Bazette's Correction (N=41) | 1
  High QTc Fredericia's Correction (N=41) | 0

14. Other Pre Specified Outcome: Adverse Events Leading to Discontinuation
Description: A listing of adverse events leading to discontinuation from the study. Abbreviation in data table: ADHD = Attention-Deficit/Hyperactivity Disorder.
Time Frame: Week 0 (Baseline) to 30 Weeks
Population: All enrolled patients.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 72
participants
  Period II/III: Nausea | 1
  Period II/III: Worsening of ADHD | 1
  Period II/III: Rash | 1
  Period IV: Irritability | 1

ADVERSE EVENTS:
Time Frame: Duloxetine - Period II/III: Week 0 (Baseline) to Week 18; Duloxetine - Period IV: Week 18 to Week 30
Description: In the opinion of the investigator, none of the Serious Adverse Events were considered related to the study drug.
Groups:
- Duloxetine - Period II/III: 20 - 120 milligrams (mg) every day, once-daily (QD), by mouth (PO) for 18 weeks; If patient is ≤40 kilograms (kg), initial dose is 20 mg, then titrated up. If patient is >40 kg, initial dose is 30 mg, then titrated up.
- Duloxetine - Period IV: 20 - 120 milligrams (mg) every day, once-daily (QD), by mouth (PO) between Weeks 18 - 30; If patient is ≤40 kilograms (kg), initial dose is 20 mg, then titrated up. If patient is >40 kg, initial dose is 30 mg, then titrated up.
Arm/Group | Duloxetine - Period II/III | Duloxetine - Period IV
Serious Adverse Events (participants affected / at risk) | 5/72 | 0/48
Other Adverse Events (participants affected / at risk) | 57/72 | 21/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine - Period II/III (N=72) | Duloxetine - Period IV (N=48)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Oppositional defiant disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine - Period II/III (N=72) | Duloxetine - Period IV (N=48)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Myopia (Eye disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (20) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (13) | 1 (1)
Fatigue (General disorders) | 5 (5) | 2 (2)
Irritability (General disorders) | 2 (2) | 1 (1)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (9) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 0 (0)
Headache (Nervous system disorders) | 10 (13) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Sedation (Nervous system disorders) | 7 (7) | 1 (1)
Somnolence (Nervous system disorders) | 7 (8) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Bruxism (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Libido increased (Psychiatric disorders) | 0 (0) | 1 (1)
Oppositional defiant disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Restlessness (Psychiatric disorders) | 2 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The Results Record was revised as a result of correcting identified errors in the number of participants with potentially significant changes in blood pressure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days